CLINICAL TRIAL: NCT03535740
Title: Brigatinib in Patients With Anaplastic Lymphoma Kinase-Positive (ALK+), Advanced Non-Small-Cell Lung Cancer (NSCLC) Progressed on Alectinib or Ceritinib
Brief Title: A Study of Brigatinib in Participants With Anaplastic Lymphoma Kinase-Positive (ALK+), Advanced Non-Small-Cell Lung Cancer (NSCLC) Progressed on Alectinib or Ceritinib
Acronym: ALTA-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ariad Pharmaceuticals (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Brigatinib-2002; 2018-000635-27 (EudraCT Number); NL66462.078.18 (Registry Identifier: CCMO); JapicCTI-194915 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-05-09; First posted 2018-05-24 (Actual); Results first posted 2021-10-25 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: ALK-positive Advanced NSCLC
Keywords: Drug Therapy
MeSH Terms: interventions — brigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Brigatinib 90 mg/180 mg With Optional Dose Escalation to 240 mg (Experimental): Brigatinib 90 mg, tablets, orally, once daily (QD) for 7 days, followed by brigatinib 180 mg, tablets, orally, QD for until objective disease progression per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, as assessed by the investigator, or intolerable toxicity. Participants who experienced progression on the 180 mg dose and had not experienced toxicities greater than Grade 2 had the option to receive brigatinib 240 mg QD based on investigator's discretion, up to 20 months until data cut-off: 30 September 2020. Participants who experienced progression on any doses but judged as still benefiting from the study treatment by the investigator may continue to use the current dose, up to study end.
  Interventions: Drug: Brigatinib

INTERVENTIONS:
Drug: Brigatinib — Brigatinib Tablets
  Other Names: AP26113

SUMMARY:
The primary purpose of this study is to determine the efficacy of brigatinib by confirmed objective response rate (ORR) by response evaluation criteria in solid tumors (Response Evaluation Criteria in Solid Tumors [RECIST]), in participants with ALK+ locally advanced or metastatic NSCLC whose disease has progressed on therapy with alectinib or ceritinib.

DETAILED DESCRIPTION:
The drug being tested in this study is called brigatinib (AP26113). Brigatinib is being tested to treat people who have anaplastic lymphoma kinase-positive (ALK+), advanced non-small-cell lung cancer (NSCLC).

The study will enroll approximately 103 patients. Participants will be assigned to the treatment group:

• Brigatinib

All participants will be asked to take brigatinib 90 mg tablet in lead-in period for 7 days, followed by brigatinib 180 mg at the same time each day throughout the study. Participants with progressive disease had an option to receive an escalated dose of brigatinib 240 mg as per investigator's discretion in case no toxicities (greater than grade 2) are experienced.

This multicenter trial will be conducted worldwide. The overall time to participate in this study is approximately 3 years. Participants will make multiple visits to the clinic, and 30 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically or cytologically confirmed stage IIIB (locally advanced or recurrent and not a participant for curative therapy) or stage IV non-small-cell lung cancer (NSCLC).
2. Must meet both of the following 2 criteria:

   1. Have documentation of anaplastic lymphoma kinase (ALK) rearrangement by a positive result from any laboratory test® approved by the food and drug administration (FDA) or Have documented ALK rearrangement by a different test (non-FDA-approved local lab tests) and have provided tumor sample to the central laboratory. (Note: Central laboratory ALK rearrangement testing results are not required to be obtained before randomization.)
   2. Had been on any one of the ALK tyrosine kinase inhibitor (TKIs) (alectinib, ceritinib, crizotinib) for at least 12 weeks before progression.
3. Had progressive disease (PD) while on alectinib or ceritinib
4. Had alectinib or ceritinib as the most recent ALK inhibitor therapy.
5. Have at least 1 measurable lesion per response evaluation criteria in solid tumors (RECIST) version 1.1 as assessed by the investigator.
6. Had recovered from toxicities related to prior anticancer therapy to national cancer institute common terminology criteria for adverse events (NCI CTCAE), version 4.03, Grade <=1. (Note: Treatment-related alopecia or peripheral neuropathy that are Grade >1 are allowed if deemed irreversible.) and have adequate major organ functions.
7. Have a life expectancy of ≥3 months.

Exclusion Criteria:

1. Had received any prior ALK-targeted TKI other than crizotinib, alectinib, or ceritinib.
2. Had received both alectinib and ceritinib.
3. Had previously received more than 3 regimens of systemic anticancer therapy for locally advanced or metastatic disease.
4. Had symptomatic brain metastasis (parenchymal or leptomeningeal). Participants with asymptomatic brain metastasis or who have stable symptoms that did not require an increased dose of corticosteroids to control symptoms in the past 7 days before the first dose of brigatinib may be enrolled.
5. Had current spinal cord compression (symptomatic or asymptomatic and detected by radiographic imaging). Participants with leptomeningeal disease and without cord compression are allowed.
6. Had a cerebrovascular accident or transient ischemic attack within 6 months before first dose of brigatinib.
7. Had an ongoing or active infection, including, but not limited to, the requirement for intravenous antibiotics.
8. Had malabsorption syndrome or other gastrointestinal (GI) illness that could affect oral absorption of brigatinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2024-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (79):
- United States (10):
  - University of California Irvine Health Chao Family Comprehensive Cancer Center, Orange, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - USOR - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Florida Hospital Medical Group, Orlando, Florida
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Levine Cancer Institute - Southpark, Charlotte, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - USOR - Virginia Cancer Specialists - Fairfax Office, Fairfax, Virginia
- Australia (3):
  - Saint Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Austria (2):
  - Klinikum Klagenfurt Am Worthersee, Klagenfurt, Carinthia
  - Krankenhaus Elisabethinen Linz, Linz, Upper Austria
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Tom Baker Cancer Center, Calgary, British Columbia
  - Toronto University Health Network, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- China (6):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Jilin Provincial Cancer Hospital (Changchun Cancer Hospital), Changchun, Jilin
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- France (5):
  - Hopital Haut-Leveque, Pessac, Aquitaine
  - Centre de Lutte Contre le Cancer Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Hopital Larrey, CHU de Toulouse, Service de Pneumologie, Toulouse, Midi-pyrenees
  - Assistance Publique-Hopitaux de Marseille Hopital Nord, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier Intercommunal de Creteil, Créteil, Île-de-France Region
- Germany (7):
  - Thoraxklinik Heidelberg gGmbH, Heidelberg, Baden-Wurttemberg
  - Universitatsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum Kempten-Oberallgau, Kempten (Allgäu), Bavaria
  - Ludwig-Maximilians-Universitat Munchen, München, Bavaria
  - Pius Hospital Oldenburg, Oldenburg, Lower Saxony
  - Evangelisches Krankenhaus Hamm, Hamm, North Rhine-Westphalia
  - HELIOS Klinikum Emil von Behring, Berlin
- Hong Kong (4):
  - Prince of Wales Hospital, Shatin, New Territories
  - Queen Mary Hospital, Hong Kong
  - Queen Elizabeth Hospital, Kowloon
  - Princess Margaret Hospital - Hong Kong, Kowloon
- Italy (7):
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Centro di Riferimento Oncologico di Aviano, Aviano, Pordenone
  - Azienda Ospedaliero - Universitaria San Luigi Gonzaga, Orbassano, Torino
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Azienda USL della Romagna, Ravenna
- Japan (6):
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Okayama University Hospital, Okayama, Okayama-ken
  - Kansai Medical University Hirakata Hospital, Hirakata-shi, Osaka
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
- Netherlands (3):
  - Maastricht University Medical Centre, Maastricht, Limburg
  - Vrije Universiteit Medisch Centrum, Amsterdam, North Holland
  - Erasmus University Medical Center, Rotterdam, South Holland
- South Korea (9):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon, Gyeonggi-do
  - Korea University Anam Hospital, Seoul, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, Gyeongsangbuk-do
  - Keimyung University Dongsan Medical Center, Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Institut Catala d'Oncologia Badalona - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Complejo Hospitalario Universitario A Coruna, A Coruña, LA Coruna
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
- Sweden (3):
  - Skanes Universitetssjukhus i Lund, Lund, Skåne County
  - Karolinska Universitetssjukhuset, Stockholm
  - Uppsala Akademiska Sjukhus, Uppsala
- Taiwan (4):
  - Changhua Christian Hospital, Changhua, Changhwa
  - National Cheng Kung University, Tainan, Tainan CITY
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Mok T, Nishio M, Yoshida T, Ahn MJ, Kudou K, Asato T, Yang H, Tong X, Vincent S, Zhang P, Yamamoto N, Kim ES. Efficacy and safety of brigatinib after alectinib in patients with ALK-positive NSCLC: Integrated analysis of the ALTA-2 and J-ALTA studies. Lung Cancer. 2025 Nov;209:108793. doi: 10.1016/j.lungcan.2025.108793. Epub 2025 Oct 9. PMID 41110382
- [Derived] Ou SI, Nishio M, Ahn MJ, Mok T, Barlesi F, Zhou C, Felip E, de Marinis F, Kim SW, Perol M, Liu G, Migliorino MR, Kim DW, Novello S, Bearz A, Garrido P, Mazieres J, Morabito A, Lin HM, Yang H, Niu H, Zhang P, Kim ES. Efficacy of Brigatinib in Patients With Advanced ALK-Positive NSCLC Who Progressed on Alectinib or Ceritinib: ALK in Lung Cancer Trial of brigAtinib-2 (ALTA-2). J Thorac Oncol. 2022 Dec;17(12):1404-1414. doi: 10.1016/j.jtho.2022.08.018. Epub 2022 Sep 10. PMID 36096442
- [Derived] Kim ES, Barlesi F, Mok T, Ahn MJ, Shen J, Zhang P, Ou SI. ALTA-2: Phase II study of brigatinib in patients with ALK-positive, advanced non-small-cell lung cancer who progressed on alectinib or ceritinib. Future Oncol. 2021 May;17(14):1709-1719. doi: 10.2217/fon-2020-1119. Epub 2021 Feb 11. PMID 33569983

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 54 investigative sites in Canada, United States, Austria, France, Germany, Italy, Netherlands, Spain, Sweden, China, Hong Kong, Japan, Korea, Taiwan, and Australia from 31 January 2019 to 21 August 2024.
Pre-assignment Details: Participants with diagnosis of ALK+, advanced NSCLC were enrolled to receive brigatinib 90 milligrams(mg) followed by 180 mg up to disease progression. 102 participants discontinued study up to interim data cut-off date: 20 May 2021. By 20 May 2021, all primary&secondary study outcome measure were met&data collection was complete. 1 participant stayed on until study completion as means to provide access to brigatinib.
Groups:
- Brigatinib 90 mg/180mg With Optional Dose Escalation to 240 mg: Participants received brigatinib 90 mg, tablets, orally, once daily (QD) for 7 days, followed by brigatinib 180 mg, tablets, orally, QD for until objective disease progression per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, as assessed by the investigator, or intolerable toxicity. Participants who experienced progression on the 180 mg dose and had not experienced toxicities greater than Grade 2 had the option to receive brigatinib 240 mg QD based on investigator's discretion, up to 28 months from start of enrollment until data cut-off: 20 May 2021.
Period: Overall Study
Arm/Group | Brigatinib 90 mg/180mg With Optional Dose Escalation to 240 mg
Started | 103
Participants Who Received Escalated Dose of Brigatinib 240 mg | 13
Completed | 0
Not Completed | 103
Not completed — Death | 44
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 13
Not completed — Site terminated by Sponsor | 45

BASELINE CHARACTERISTICS:
Population: Full Analysis Population included all participants who received at least 1 dose of brigatinib.
Groups:
- Brigatinib 90 mg/180 mg With Optional Dose Escalation to 240 mg: Participants received brigatinib 90 mg, tablets, orally, QD for 7 days, followed by brigatinib 180 mg, tablets, orally, QD for until objective disease progression per RECIST version 1.1, as assessed by the investigator, or intolerable toxicity. Participants who experienced progression on the 180 mg dose and had not experienced toxicities greater than Grade 2 had the option to receive brigatinib 240 mg QD based on investigator's discretion, up to 28 months from start of enrollment until data cut-off: 20 May 2021.
Arm/Group | Brigatinib 90 mg/180 mg With Optional Dose Escalation to 240 mg
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 92
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 49
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 44
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 6
  United States | 7
  Austria | 1
  France | 7
  Germany | 3
  Italy | 16
  Netherlands | 2
  Spain | 11
  Sweden | 2
  China | 14
  Hong Kong | 6
  Japan | 3
  Korea, South | 20
  Taiwan, Province Of China | 4
  Australia | 1
Weight [Mean (Standard Deviation); unit: kilograms (kg)] — Population: Number analyzed signifies the number of participants with data available for weight.
  kilograms (kg)
    number analyzed (Participants) | 102
    (all) | 69.23 (15.409)
Height [Mean (Standard Deviation); unit: centimeters (cm)] — Population: Number analyzed signifies the number of participants with data available for height.
  centimeters (cm)
    number analyzed (Participants) | 100
    (all) | 165.86 (10.172)

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (ORR) Using RECIST v1.1 as Assessed by the Independent Review Committee (IRC)
Description: Confirmed ORR is defined as the percentage of the participants who are confirmed to have achieved complete response (CR) or partial response (PR), per RECIST version 1.1 (confirmed ≥4 weeks after initial response), after the initiation of study treatment. CR: disappearance of all extranodal target lesions and all pathological lymph nodes must have decreased to <10 mm in short axis and PR: at least a 30% decrease in the sum of the longest diameters (SLD) of target lesions taking as reference the Baseline sum diameters. Percentages were rounded off to the nearest single decimal place.
Time Frame: Up to approximately 20 months from the start of enrollment till data cut-off 30 September 2020
Population: Full Analysis Population included all participants who received at least 1 dose of brigatinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brigatinib 90 mg/180 mg With Optional Dose Escalation to 240 mg
Number analyzed (Participants) | 103
percentage of participants | 26.2 [18.0 to 35.8]
Statistical Analysis 1: Comparison: Brigatinib 90 mg/180 mg With Optional Dose Escalation to 240 mg; Test type: Other; p = 0.0763, Exact Binomial Test — P-value was based on the comparison of the confirm ORR among the 90/180mg group against a fixed response rate of 20%; The calculation was based on an exact binomial test with a total 1-sided alpha level of 0.025 at primary analysis

2. Secondary Outcome: Confirmed ORR Using RECIST v1.1 as Assessed by the Investigator
Description: Confirmed ORR is defined as the percentage of the participants who are confirmed to have achieved CR or PR, per RECIST version 1.1 (confirmed ≥4 weeks after initial response), after the initiation of study treatment. CR: disappearance of all extranodal target lesions and all pathological lymph nodes must have decreased to <10 mm in short axis and PR: at least a 30% decrease in the SLD of target lesions taking as reference the baseline sum diameters. Percentages were rounded off to the nearest single decimal place.
Time Frame: Up to approximately 28 months
Population: Full Analysis Population included all participants who received at least 1 dose of brigatinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brigatinib 90 mg/180 mg With Optional Dose Escalation to 240 mg
Number analyzed (Participants) | 103
percentage of participants | 26.2 [18.0 to 35.8]

3. Secondary Outcome: Duration of Response (DOR) as Assessed by the IRC and the Investigator
Description: DOR is defined as the time interval from the time that the measurement criteria are first met for CR or PR until the first date that the progressive disease (PD) is objectively documented, or death. CR: disappearance of all extranodal target lesions and all pathological lymph nodes must have decreased to <10 mm in short axis. PR: at least a 30% decrease in the SLD of target lesions taking as reference the Baseline sum diameters. PD: SLD increased by at least 20% from the smallest value on study (including Baseline, if that is the smallest). SLD must also demonstrate an absolute increase of at least 5 mm (2 lesions increasing from, for example, 2 mm to 3 mm, does not qualify).
Time Frame: Up to approximately 28 months
Population: Full Analysis Population included all participants who received at least 1 dose of brigatinib. Overall number of participants analyzed is the number of participants who were responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 90 mg/180 mg With Optional Dose Escalation to 240 mg
Number analyzed (Participants) | 27
months
  IRC-Assessed DOR | 6.341 [5.552 to NA] — The upper limit of 95 % confidence interval was not estimable due to insufficient number of events observed among the responding participants.
  Investigator-Assessed DOR | 6.735 [4.435 to 9.232]

4. Secondary Outcome: Progression-Free Survival (PFS) as Assessed by the IRC and the Investigator
Description: PFS is defined as the time interval from the date of the first dose of the study treatment until the first date at which disease progression is objectively documented, or death due to any cause, whichever occurs first. PFS was censored for participants without documented disease progression or death.
Time Frame: Up to approximately 28 Months
Population: Full Analysis Population included all participants who received at least 1 dose of brigatinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 90 mg/180 mg With Optional Dose Escalation to 240 mg
Number analyzed (Participants) | 103
months
  IRC-Assessed PFS | 3.811 [3.515 to 5.848]
  Investigator-Assessed PFS | 3.811 [3.154 to 5.552]

5. Secondary Outcome: Disease Control Rate (DCR) as Assessed by the IRC and the Investigator
Description: DCR is defined as the percentage of participants who have achieved CR, PR or stable disease (SD) (in the case of SD, measurements must have met the SD criteria at least once after study entry at a minimum interval of 6 weeks) after the initiation of study treatment. CR: disappearance of all extranodal target lesions and all pathological lymph nodes must have decreased to <10 mm in short axis. PR: at least a 30% decrease in the SLD of target lesions taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Percentages were rounded off to the nearest single decimal place.
Time Frame: Up to approximately 28 months
Population: Full Analysis Population included all participants who received at least 1 dose of brigatinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brigatinib 90 mg/180 mg With Optional Dose Escalation to 240 mg
Number analyzed (Participants) | 103
percentage of participants
  IRC-Assessed DCR | 54.4 [44.3 to 64.2]
  Investigator-Assessed DCR | 59.2 [49.1 to 68.8]

6. Secondary Outcome: Time to Response as Assessed by the IRC and the Investigator
Description: Time to response is defined as the time interval from the date of the first dose of the study treatment until the initial observation of CR or PR. CR: disappearance of all extranodal target lesions and all pathological lymph nodes must have decreased to <10 mm in short axis. PR: at least a 30% decrease in the SLD of target lesions taking as reference the baseline sum diameters.
Time Frame: Up to approximately 28 months
Population: as for outcome 3
Measure: Median (Full Range); unit: months
Arm/Group | Brigatinib 90 mg/180 mg With Optional Dose Escalation to 240 mg
Number analyzed (Participants) | 27
months
  IRC-Assessed Time to Response | 1.807 [1.45 to 5.36]
  Investigator-Assessed Time to Response | 1.807 [1.58 to 10.87]

7. Secondary Outcome: Confirmed Intracranial Objective Response Rate (iORR) in Participants With Brain Metastases at Baseline, as Assessed by the IRC
Description: Confirmed iORR is defined as the percentage of the participants who have achieved CR or PR in the brain per a modification of RECIST version 1.1, after the initiation of study treatment, in participants with intracranial brain metastases at baseline. CR: disappearance of all extranodal target lesions and all pathological lymph nodes must have decreased to <10 mm in short axis. or partial response or PR: at least a 30% decrease in the SLD of target lesions taking as reference the baseline sum diameters. Percentages were rounded off to the nearest single decimal place.
Time Frame: Up to approximately 28 months
Population: Intracranial central nervous system (iCNS) disease population included those participants in the Full Analysis Population who were determined by the IRC to have iCNS metastases at baseline, regardless of whether they had at least 1 lesion that qualified as a target lesion in their baseline assessment by the IRC.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brigatinib 90 mg/180 mg With Optional Dose Escalation to 240 mg
Number analyzed (Participants) | 55
percentage of participants | 14.5 [6.5 to 26.7]

8. Secondary Outcome: Duration of Intracranial Response in Participants With Brain Metastases at Baseline, as Assessed by the IRC
Description: Duration of intracranial response is defined as the time interval from the time that the measurement criteria are first met for CR or PR until the first date that PD (including baseline, if that is the smallest). SLD must also demonstrate an absolute increase of at least 5 mm. (2 lesions increasing from, for example, 2 mm to 3 mm, does not qualify) in the brain is objectively documented or death, in participants with intracranial metastases at baseline. CR: disappearance of all extranodal target lesions and all pathological lymph nodes must have decreased to <10 mm in short axis. or partial response or PR: at least a 30% decrease in the SLD of target lesions taking as reference the baseline sum diameters in the brain. PD: SLD increased by at least 20% from the smallest value on study.
Time Frame: Up to approximately 28 months
Population: iCNS disease population included those participants in the Full Analysis Population who were determined by the IRC to have iCNS metastases at baseline, regardless of whether they had at least 1 lesion that qualified as a target lesion in their baseline assessment by the IRC. Overall number of participants analyzed is the number of participants who were responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 90 mg/180 mg With Optional Dose Escalation to 240 mg
Number analyzed (Participants) | 8
months | NA [5.717 to NA] — The median and upper limit of 95 % confidence interval was not estimable due to insufficient number of events observed among the responding participants.

9. Secondary Outcome: Intracranial Progression-Free Survival (iPFS) in Participants With Brain Metastases at Baseline, as Assessed by the IRC
Description: iPFS is defined as the time interval from the date of the first dose of the study treatment until the first date at which intracranial brain disease progression is objectively documented, or death due to any cause, whichever occurs first, in participants with intracranial metastases at enrollment. iPFS will be censored for participants without documented intracranial disease progression or death.
Time Frame: Up to approximately 28 months
Population: iCNS disease population included of those participants in the Full Analysis Population who were determined by the IRC to have iCNS metastases at baseline, regardless of whether they had at least 1 lesion that qualified as a target lesion in their baseline assessment by the IRC.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 90 mg/180 mg With Optional Dose Escalation to 240 mg
Number analyzed (Participants) | 55
months | 5.224 [3.515 to 7.392]

10. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time interval from the date of the first dose of the study treatment until death due to any cause. It was censored on the date of last contact for those participants who were alive.
Time Frame: Up to approximately 28 months
Population: Full Analysis Population included all participants who received at least 1 dose of brigatinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 90 mg/180 mg With Optional Dose Escalation to 240 mg
Number analyzed (Participants) | 103
months | 21.290 [12.189 to NA] — The upper limit of 95 % confidence interval was not estimable due to insufficient number of events observed among the responding participants.

11. Secondary Outcome: Number of Participants With One or More Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. This includes any newly occurring event, or a previous condition that has increased in severity or frequency since the administration of study drug. TEAE: any AE either reported for the first time or worsening of a pre-existing event after first dose of study drug and within 30 days of the last administration of study drug.
Time Frame: First dose of study drug up to 30 days after last dose (approximately 5 years)
Population: Safety Analysis Population included all participants who received at least 1 dose of brigatinib. As pre-specified in protocol, AEs are reported for 2 sets/arms. Arm 1 (brigatinib 90/180 mg) and Arm 2 (brigatinib 240 mg).
Measure: Count of Participants; unit: Participants
Groups:
- Brigatinib 90/180 mg: Brigatinib 90 mg, tablets, orally, QD for 7 days, followed by Brigatinib 180 mg, tablets, orally, QD for until objective disease progression per RECIST version 1.1, as assessed by the investigator, or intolerable toxicity up to approximately 28 months from start of enrollment till data cut-off: 20 May 2021. Participants who experienced progression on any doses but judged as still benefiting from the study treatment by the investigator continued to use the current dose, up to study end.
- Brigatinib 240 mg: Participants who experienced progression on the 180 mg dose and had not experienced toxicities greater than Grade 2 had the option to receive brigatinib 240 mg QD from start of enrollment based on investigator's discretion up to data-cut off: 20 May 2021 (approximately 28 months). Participants who experienced progression on any doses but judged as still benefiting from the study treatment by the investigator continued to use the current dose, up to study end.
Arm/Group | Brigatinib 90/180 mg | Brigatinib 240 mg
Number analyzed (Participants) | 103 | 13
Participants | 103 | 12

12. Secondary Outcome: Number of Participants With Improvement in Health-Related Quality of Life (HRQOL) Based on European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Score
Description: EORTC QLQ-C30 incorporates 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). EORTC QLQ-C30 contains 28 questions (4-point scale where 1=Not at all [best] to 4=Very Much [worst]) and 2 questions (7-point scale where 1=Very poor [worst] to 7= Excellent [best]). Raw scores are converted into scale scores ranging from 0 to 100. For the functional scales and the global health status scale, higher scores represent better quality of life (QOL); for the symptom scales, lower scores represent better QOL. Improvement is defined as a change from baseline of 10 or more points higher for functional scales and 10 or more points lower for symptom scales.
Time Frame: Up to approximately 28 months
Population: Full Analysis Population included all participants who received at least 1 dose of brigatinib. Overall number of participants analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis for the specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Brigatinib 90 mg/180 mg With Optional Dose Escalation to 240 mg
Number analyzed (Participants) | 93
Participants
  Global Health Status/QoL | 52
  Physical Functioning | 55
  Role Functioning | 53
  Emotional Functioning | 36
  Cognitive Functioning | 47
  Social Functioning | 53
  Fatigue | 55
  Nausea and Vomiting | 21
  Pain | 48
  Dyspnoea Raw | 26
  Insomnia | 40
  Appetite Loss | 30
  Constipation: number analyzed (Participants) | 92
  Constipation | 23
  Diarrhoea | 27
  Financial Difficulties | 27

13. Secondary Outcome: Number of Participants With Improvement of HRQOL Based on EORTC QLQ- Lung Cancer (LC) 13
Description: HRQOL scores will be assessed with EORTC, its lung cancer module QLQ-LC13. QLQ-LC13 contains 13 questions assessing lung cancer-associated symptoms (cough, hemoptysis, dyspnea, and site-specific pain), treatment-related side effects (sore mouth, dysphagia, peripheral neuropathy, and alopecia), and use of pain medication. Scale score range: 0 to 100. Higher symptom score = greater degree of symptom severity. Improvement is defined as a change from baseline of 10 or more points lower for symptom scales.
Time Frame: Up to approximately 28 months
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Brigatinib 90 mg/180 mg With Optional Dose Escalation to 240 mg
Number analyzed (Participants) | 93
Participants
  Composite Endpoint Score | 61
  Dyspnoea | 45
  Coughing | 37
  Haemoptysis | 4
  Sore Mouth | 6
  Dysphagia | 4
  Peripheral Neuropathy | 25
  Alopecia | 14
  Pain in Chest | 24
  Pain in Arm or Shoulder | 23
  Pain in Other Parts: number analyzed (Participants) | 92
  Pain in Other Parts | 41

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 30 days after last dose (approximately 5 years)
Description: Safety Analysis Population: participants who received at least 1 dose of brigatinib. As pre-specified in protocol all-cause mortality and AEs are reported separately for 2 sets/arms: Arm 1 (brigatinib 90/180 mg) and Arm 2 (brigatinib 240 mg).
Groups:
- Brigatinib 90/180 mg: Participants received brigatinib 90 mg, tablets, orally, QD for 7 days, followed by brigatinib 180 mg, tablets, orally, QD for until objective disease progression per RECIST version 1.1, as assessed by the investigator, or intolerable toxicity. Participants who experienced progression on the 180 mg dose and had not experienced toxicities greater than Grade 2 had the option to receive brigatinib 240 mg QD based on investigator's discretion, up to 28 months from start of enrollment until data cut-off: 20 May 2021.
- Brigatinib 240 mg: Participants who experienced progression on the 180 mg dose and had not experienced toxicities greater than Grade 2 had the option to receive brigatinib 240 mg QD from start of enrolment based on investigator's discretion up to data-cut off: 30 September 2020 (approximately 20 months). Participants who experienced progression on any doses but judged as still benefiting from the study treatment by the investigator may continue to use the current dose, up to study end.
Arm/Group | Brigatinib 90/180 mg | Brigatinib 240 mg
All-Cause Mortality (participants affected / at risk) | 39/103 | 5/13
Serious Adverse Events (participants affected / at risk) | 48/103 | 3/13
Other Adverse Events (participants affected / at risk) | 98/103 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brigatinib 90/180 mg (N=103) | Brigatinib 240 mg (N=13)
Abdominal sepsis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 0
Complication of device insertion (General disorders) | 1 | 0
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 | 0
Death (General disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Disease progression (General disorders) | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hospitalisation (Surgical and medical procedures) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Meningitis (Infections and infestations) | 1 | 0
Metastases to biliary tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Moyamoya disease (Nervous system disorders) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pain (General disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 3 | 0
Sepsis (Infections and infestations) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brigatinib 90/180 mg (N=103) | Brigatinib 240 mg (N=13)
Abdominal pain upper (Gastrointestinal disorders) | 6 | 0
Alanine aminotransferase increased (Investigations) | 19 | 2
Amylase increased (Investigations) | 16 | 2
Anaemia (Blood and lymphatic system disorders) | 10 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 6 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 1
Aspartate aminotransferase increased (Investigations) | 22 | 3
Asthenia (General disorders) | 13 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 0
Blood alkaline phosphatase increased (Investigations) | 9 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Blood calcium increased (Investigations) | 2 | 1
Blood cholesterol increased (Investigations) | 5 | 2
Blood creatine phosphokinase increased (Investigations) | 35 | 5
Blood creatinine increased (Investigations) | 5 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Chest pain (General disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 11 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 3
Cytokine release syndrome (Immune system disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 11 | 1
Diarrhoea (Gastrointestinal disorders) | 41 | 7
Dizziness (Nervous system disorders) | 10 | 0
Dysgeusia (Nervous system disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Fatigue (General disorders) | 4 | 1
Gamma-glutamyltransferase increased (Investigations) | 8 | 0
Headache (Nervous system disorders) | 16 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 1
Hypertension (Vascular disorders) | 20 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 1
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 3 | 1
Lipase increased (Investigations) | 19 | 1
Localised infection (Infections and infestations) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Mucosal inflammation (General disorders) | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 1
Nausea (Gastrointestinal disorders) | 29 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 8 | 0
Oedema peripheral (General disorders) | 8 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 0
Paraesthesia (Nervous system disorders) | 4 | 1
Persistent depressive disorder (Psychiatric disorders) | 0 | 1
Platelet count decreased (Investigations) | 3 | 1
Pneumonia (Infections and infestations) | 8 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1
Pyrexia (General disorders) | 13 | 2
Rash (Skin and subcutaneous tissue disorders) | 8 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (General disorders) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Tunnel vision (Nervous system disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 18 | 2
Weight decreased (Investigations) | 14 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT03535740/Prot_002.pdf
  • Statistical Analysis Plan (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT03535740/SAP_001.pdf